CLINICAL TRIAL: NCT03140566
Title: Ultrasound Evaluation of the Inferior Vena Cava in Addition to Clinical Assessment to Guide Decongestion in Acute Decompensated Heart Failure: a Pilot Study
Brief Title: Ultrasound Evaluation of the IVC in Addition to Clinical Assessment to Guide Decongestion in ADHF
Acronym: CAVA-ADHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Holger Thiele, Director, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAVA-ADHF-DZHK10
Record Dates: First submitted 2017-04-25; First posted 2017-05-04 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure
Keywords: heart failure; acute decompensated heart failure; congestion; inferior vena cava
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical assessment plus IVC diameter (Experimental): Decongesting treatment guided by clinical assessment and ultrasound evaluation of the inferior vena cava diameter
  Interventions: Diagnostic Test: Ultrasound evaluation of the inferior vena cava diameter
- Clinical assessment only (Sham Comparator): Decongesting treatment guided by clinical assessment alone
  Interventions: Diagnostic Test: Sham ultrasound evaluation of the inferior vena cava diameter

INTERVENTIONS:
Diagnostic Test: Ultrasound evaluation of the inferior vena cava diameter — Treatment will be guided by clinical assessment and ultrasound evaluation of the inferior vena cava (IVC) diameter. Decongestion should lead to maximal IVC diameter ≤2.1 cm and IVC collapsibility index >50% in addition to relief of symptoms and signs of congestion before discharge.
  Arms: Clinical assessment plus IVC diameter
Diagnostic Test: Sham ultrasound evaluation of the inferior vena cava diameter — Teatment guided by clinical assessment alone. Decongestion should lead to relief of symptoms and signs of congestion before discharge. IVC ultrasound evaluation is performed, but results are not reported to treating physicians.
  Arms: Clinical assessment only

SUMMARY:
CAVA-ADHF is designed as a prospective, randomized, controlled, patient-blinded, multicenter, parallel-group trial. The objective is to test whether evaluation of the inferior vena cava diameter in addition to clinical assessment is superior compared to clinical assessment alone with respect to the surrogate endpoint of change in NT-proBNP from baseline to discharge. The CAVA-ADHF trial is supported by the Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK).

DETAILED DESCRIPTION:
Only limited evidence is available on the best method to monitor and guide decongestion in acute decompensated heart failure. Therefore, no specific guideline recommendations are made in this regard. It is unknown whether an objective congestion marker can be used to guide decongestion or such marker is only of prognostic value by identifying high-risk patients with an advanced disease state.

CAVA-ADHF is designed as prospective, randomized, controlled, patient-blinded, multicenter, parallel-group trial and aims to demonstrate effectiveness of inferior vena cava (IVC)-guided decongestion, its feasibility, and to estimate effect size and variability of clinical endpoints following the intention-to-treat principle.

After inclusion and exclusion criteria have been checked patients will be randomized:

Experimental intervention: Decongesting treatment guided by clinical assessment and ultrasound evaluation of the IVC diameter. Decongestion should lead to a maximal IVC diameter ≤2.1 cm and IVC collapsibility index >50% in addition to relief of symptoms and signs of congestion before discharge.

Control intervention: Decongesting treatment guided by clinical assessment alone. The IVC ultrasound evaluation is performed, but results are not reported to treating physicians.

Trial intervention will end with discharge from the index hospitalization. Patients will be followed-up for 180 to 210 days after randomization.

The CAVA-ADHF trial is supported by the Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for ADHF with dyspnea ≥NYHA III, peripheral edema, and pulmonary congestion (rales on auscultation or pulmonary vascular congestion on chest radiograph)
* Age ≥18 years
* NT-proBNP >300 ng/l within 24 h after admission
* Sufficient ultrasound visualization to evaluate IVC
* IVCmax >2.1 cm and IVCCI ≤50 % in the baseline assessment within 24 h after admission
* Capability to sign informed consent personally

Exclusion Criteria:

* Cardiogenic shock with systolic blood pressure <90 mmHg plus end-organ hypoperfusion
* ADHF due to significant arrhythmias
* Severe pulmonary disease as primary cause of dyspnea
* Simplified Modification of Diet in Renal Disease estimated glomerular filtration rate <30 ml/min/1.73 m²
* Need for non-invasive or invasive ventilation support at baseline
* Pregnancy
* Participation in another interventional trial regarding heart failure treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2017-06-03 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Change in NT-proBNP from baseline to discharge | Measured at baseline (within 24 hours of admission to index hospitalization) and on the day of discharge from index hospitalization (discharge planning is at the discretion of treating physician but will be around 5 to 8 days after admission)
  The core laboratory at Luebeck will determine NT-proBNP levels for calculation of the endpoint from samples obtained at baseline and at discharge.

SECONDARY OUTCOMES:
Proportion of patients with IVC ultrasound on two thirds of days in hospital and at discharge among all randomized patients | Measured on the day of discharge from index hospitalization (discharge planning is at the discretion of treating physician but will be around 5 to 8 days after admission)
  Proportion of patients with per-protocol treatment in the experimental group.
All-cause mortality | 180 days after randomization
  Participants will be contacted by telephone at 180 days (180 to 210 days) after randomization to assess vital status (all-cause mortality). In case of unavailability patients, relatives, general practitioners, and/or population register will be contacted.
Cardiovascular mortality | 180 days after randomization
  Participants will be contacted by telephone at 180 days (180 to 210 days) after randomization to assess vital status (all-cause mortality). In case of unavailability patients, relatives, general practitioners, and/or population register will be contacted. Medical reports will be requested to adjudicate cause of death.
Unscheduled readmission for any cause | 180 days after randomization
  Participants will be contacted by telephone at 180 days (180 to 210 days) after randomization to assess readmission status. In case of unavailability patients, relatives, general practitioners, and/or population register will be contacted.
Readmission for heart failure | 180 days after randomization
  Participants will be contacted by telephone at 180 days (180 to 210 days) after randomization to assess readmission status. In case of unavailability patients, relatives, general practitioners, and/or population register will be contacted. Medical reports will be requested to adjudicate cause of readmission.
Hemoconcentration | Measured at baseline (within 24 hours of admission to index hospitalization) and on the day of discharge from index hospitalization (discharge planning is at the discretion of treating physician but will be around 5 to 8 days after admission)
  Hemoconcentration will be defined as a relative increase in hemoglobin from baseline to discharge.
Freedom from signs of congestion at discharge | Measured on the day of discharge from index hospitalization (discharge planning is at the discretion of treating physician but will be around 5 to 8 days after admission)
  Freedom from signs of congestion at discharge is defined as the absence of orthopnea, pulmonary rales, and jugular venous distension in conjunction with none or only a trace of edema at discharge.
Cumulative loop diuretic dose during index hospitalization | Measured on the day of discharge from index hospitalization (discharge planning is at the discretion of treating physician but will be around 5 to 8 days after admission)
  For calculation of the cumulative loop diuretic dose during index hospitalization all intrahospital applied doses of loop diuretics will be converted to intravenous furosemide equivalents and summed up. Preclinical doses applied by the emergency medical services will not be considered.
Length of index hospitalization | Measured on the day of discharge from index hospitalization (discharge planning is at the discretion of treating physician but will be around 5 to 8 days after admission)
  Time in days from hospital admission to hospital dicharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitäres Herzzentrum Lübeck, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jobs A, Rausch TK, Konig IR, Vonthein R, Devendra A, Schafer J, Nauck M, Eitel I, Stiermaier T, Laugwitz KL, Ledwoch J, Valentova M, von Haehling S, Stork S, Arnold N, Karakas M, Westermann D, Lenz T, Gori T, Edelmann F, Seppelt P, Felix SB, Lutz M, Hedwig F, Akin I, Scherer C, Desch S, Thiele H; CAVA-ADHF-DZHK10 Investigators. Inferior Vena Cava Ultrasound to Guide Decongestion in Acute Decompensated Heart Failure: A Randomized Controlled Trial. JACC Heart Fail. 2025 Oct;13(10):102578. doi: 10.1016/j.jchf.2025.102578. Epub 2025 Sep 9. PMID 40929999